CLINICAL TRIAL: NCT06821750
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO CONTROLLED, DOSE ESCALATING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF SINGLE AND MULTIPLE SUBCUTANEOUS DOSES OF PF-07314470 IN HEALTHY PARTICIPANTS
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-07314470 Are Tolerated and Act in the Body in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor has decided to terminate the above referenced clinical study for business reasons. There were no safety concerns that led to this decision and there was no impact to participant safety.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: C5271001
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- PF-07314470; Cohorts 1 to 7, optional Cohort 8 and optional Japanese Cohort 14 (Experimental): Participants will receive a single dose of PF-07314470 at 1 of 7 dose levels
  Interventions: Biological: PF-07314470
- Placebo for PF-07314470; Cohorts 1 to 7, optional Cohort 8 and optional Japanese Cohort 14 (Placebo Comparator): Participants will receive a single dose of placebo for PF-07314470
  Interventions: Biological: Placebo for PF-07314470
- PF-07314470; Cohorts 9 to 13 (Experimental): Participants will receive PF-07314470 weekly at 1 of 4 dose levels for 4 doses, or every 2 weeks at 1 dose level for 3 doses.
  Interventions: Biological: PF-07314470
- Placebo for PF-07314470; Cohorts 9 to 13 (Placebo Comparator): Participants will receive placebo for PF-07314470 weekly for 4 doses, or every 2 weeks for 3 doses.
  Interventions: Biological: Placebo for PF-07314470

INTERVENTIONS:
Biological: PF-07314470 — subcutaneous injection
  Arms: PF-07314470; Cohorts 1 to 7, optional Cohort 8 and optional Japanese Cohort 14; PF-07314470; Cohorts 9 to 13
Biological: Placebo for PF-07314470 — subcutaneous injection
  Arms: Placebo for PF-07314470; Cohorts 1 to 7, optional Cohort 8 and optional Japanese Cohort 14; Placebo for PF-07314470; Cohorts 9 to 13

SUMMARY:
The purpose of this clinical trial is to learn if the study medicine (called PF-07314470) is safe and how it gets in and out of the body in healthy people.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy males aged 18 to 45 years and healthy females aged 18 to 55 years
* Body Mass Index (BMI) of 16-32 kg/m2, and a total body weight greater than 50 kg (110 lb); for Japanese participants only, a total body weight greater than 45 kg
* for Japanese participants only, enrolling as Japanese must have 4 biological grandparents who were born in Japan.

Key Exclusion Criteria:

* Evidence or history of clinically significant medical or psychiatric conditions
* Prior or current use of any prohibited medications
* History of alcohol abuse or repeated binge drinking and/or any other illicit drug use or dependence within 6 months of screening
* Pregnant or breastfeeding females, males with partners currently pregnant, or males or females pursuing artificial reproductive technologies
* Use of tobacco/nicotine containing products

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events Following Single Doses | Day 1 up to approximately Day 35
Number of Participants with Clinically Significant Change from Baseline in Laboratory Values Following Single Doses | Baseline up to approximately Day 35
Number of Participants with Clinically Significant Change from Baseline in Vital Signs Following Single Doses | Baseline up to approximately Day 35
Number of Participants with Clinically Significant Change from Baseline in ECGs Following Single Doses | Baseline up to approximately Day 35
Number of Participants with Treatment Emergent Adverse Events Following Multiple Doses | Day 1 up to approximately Day 64
Number of Participants with Clinically Significant Change from Baseline in Laboratory Values Following Multiple Doses | Baseline up to approximately Day 64
Number of Participants with Clinically Significant Change from Baseline in Vital Signs Following Multiple Doses | Baseline up to approximately Day 64
Number of Participants with Clinically Significant Change from Baseline in ECGs Following Multiple Doses | Baseline up to approximately Day 64
Number of Participants with Serious Adverse Events Following Single Doses | Day 1 up to approximately Day 35
Number of Participants with Serious Adverse Events Following Multiple Doses | Day 1 up to approximately Day 64

SECONDARY OUTCOMES:
Area Under the Serum Concentration-time Curve from Time Zero to Time of Last Measurable Concentration (AUClast) of PF-07314470 Following Single Doses | Day 1 up to approximately Day 35
Maximum Observed Serum Concentration (Cmax) of PF-07314470 Following Single Doses | Day 1 up to approximately Day 35
Time to Reach Maximum Observed Serum Concentration (Tmax) of PF-07314470 Following Single Doses | Day 1 up to approximately Day 35
Area Under the Serum Concentration-time Curve from Time Zero to Extrapolated Infinite Time (AUCinf) of PF-07314470 Following Single Doses | Day 1 up to approximately Day 35
  If data permit
Terminal Serum Elimination Half-life (t 1/2) of PF-07314470 Following Single Doses | Day 1 up to approximately Day 35
  If data permit
Area Under the Serum Concentration-time Curve at Steady State Over the Dosing Interval (AUCtau) of PF-07314470 Following Multiple Doses | Day 1 up to approximately Day 64
Maximum Observed Serum Concentration (Cmax) of PF-07314470 Following Multiple Doses | Day 1 up to approximately Day 64
Time to Reach Maximum Observed Serum Concentration (Tmax) of PF-07314470 Following Multiple Doses | Day 1 up to approximately Day 64
Terminal Serum Elimination Half-life (t 1/2) of PF-07314470 Following Multiple Doses | Day 1 up to approximately Day 64
  If data permit
Incidence of the Development of Antidrug Antibodies Against PF-07314470 Following Single Doses | Day 1 up to approximately Day 35
Incidence of the Development of Neutralizing Antibodies Against PF-07314470 Following Single Doses | Day up to approximately Day 35
  If appropriate
Incidence of the Development of Antidrug Antibodies Against PF-07314470 Following Multiple Doses | Day 1 up to approximately Day 64
Incidence of the Development of Neutralizing Antibodies Against PF-07314470 Following Multiple Doses | Day 1 up to approximately Day 64
  If appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5271001